CLINICAL TRIAL: NCT07245368
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Single Ascending and Multiple Ascending Dose Study Investigating PRA-216 in Healthy Volunteers Followed by a Phase 2a Randomized, Double-Blind, Placebo-Controlled Study in Participants With Mild-to-Moderate Asthma
Brief Title: Study of PRA-216 in Healthy Participants and Participants With Mild-to-Moderate Asthma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prana Therapies Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRA-216-101
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Mild to Moderate Asthma
Keywords: healthy volunteers; pharmacodynamics; immunogenicity; asthma; pharmacokinetics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Phase 1, Part 1: SAD Cohorts: Active Drug (Experimental): Healthy volunteers will receive a single dose of PRA-216 in a dose escalation format.
  Interventions: Drug: PRA-216
- Phase 1, Part 1: SAD Cohorts: Placebo (Placebo Comparator): Healthy volunteers will receive a single dose of placebo
  Interventions: Drug: Placebo
- Phase 1, Part 2: MAD Cohort: Active Drug (Experimental): Healthy volunteers will receive repeated doses of PRA-216 in a dose escalation format.
  Interventions: Drug: PRA-216
- Phase 1, Part 2 MAD Cohort: Placebo Comparator (Placebo Comparator): Healthy volunteers will receive repeated doses of placebo comparator.
  Interventions: Drug: Placebo
- Phase 2a: Participants with mild to moderate asthma-active drug (Experimental): Participants with mild to moderate asthma will be randomized to receive repeat doses of PRA-216.
  Interventions: Drug: PRA-216
- Phase 2a: Participants with mild to moderate asthma-placebo (Placebo Comparator): Participants with mild to moderate asthma will be randomized to receive repeat doses of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRA-216 — biologic
  Arms: Phase 1, Part 1: SAD Cohorts: Active Drug; Phase 1, Part 2: MAD Cohort: Active Drug; Phase 2a: Participants with mild to moderate asthma-active drug
Drug: Placebo — matching placebo for PRA-216
  Arms: Phase 1, Part 1: SAD Cohorts: Placebo; Phase 1, Part 2 MAD Cohort: Placebo Comparator; Phase 2a: Participants with mild to moderate asthma-placebo

SUMMARY:
Phase 1 of this study will consist of 2 parts

* Part 1 will evaluate the safety, tolerability, pharmacokinetics and immunogenicity of PRA-216 in healthy volunteers through single ascending dose administered by either intravenous (IV) or subcutaneous (SC).
* Part 2 will evaluate the safety, tolerability, pharmacokinetics (PK) and immunogenicity of PRA-216 in healthy volunteers with repeat doses of multiple ascending dose administered subcutaneously.

Phase 2a of this study is a randomized, double-blind, placebo-controlled study to investigate the efficacy, safety and immunogenicity of PRA-216 in participants with mild to moderate asthma. The dose of PRA-216 for this phase will be determined from Phase 1.

DETAILED DESCRIPTION:
This study is a Phase 1/2a randomized, double-blind, placebo-controlled, single- and multiple-dose study with staggered dose escalations in healthy participants and participants with mild to moderate asthma. Single-ascending dose (SAD) cohorts will be evaluated for one single dose administered. Multiple ascending dose (MAD) cohorts will be evaluated for repeat doses .

Participants with mild to moderate asthma will be recruited for Phase 2a of this study, to evaluate safety of randomized, double blind, placebo controlled PRA-216. The dose of PRA-216 for this phase will be determined from Phase 1 safety, tolerability, and PK data. Additional dose levels or schedules may be used for Phase 2a, depending on data from Phase 1.

This study consists of 2 phases, as follows:

Phase 1, Part 1:

SAD in healthy volunteers. Study visits in this section will entail a single dose administration of PRA-216 or placebo and collection of study data.

Phase 1, Part 2:

MAD in healthy volunteers. Study visits in this section will entail repeat doses of PRA-216 or placebo and collection of study data.

Phase 2a Participants with mild to moderate asthma will receive PRA-216 or placebo. The dose will be determined from Phase 1.

ELIGIBILITY:
Phase 1

Inclusion Criteria:

* Age 18-65
* Must be in good health with no significant medical history
* Willing and able to attend all study visits, comply with study requirements
* Able and willing to provide written informed consent

Exclusion Criteria:

* Evidence of clinically significant condition or disease
* Any physical or psychological condition that prohibits study completion
* Known history of illicit drug use or drug abuse, harmful alcohol use (at the Investigator's discretion), alcoholism, and/or smoking or nicotine-containing product use within 3 months prior to the first dose of study agent
* History of severe allergic reactions or hypersensitivity
* Donation or loss of ≥ 1 unit of whole blood or plasma within 2 months prior to dosing

Phase 2a

Inclusion criteria:

* Age 18-65
* Must be in good health with no significant medical history
* Willing and able to attend all study visits, comply with study requirements.
* Able and willing to provide written informed consent
* Documented asthma diagnosis prior for at least 12 months prior to screening.
* Symptomatic asthma
* Currently receiving maintenance asthma medications

Exclusion Criteria:

* Evidence of clinically significant condition or disease
* Known history of illicit drug use or drug abuse, harmful alcohol use (at the Investigator's discretion), alcoholism, and/or smoking or nicotine-containing product use within 3 months prior to the first dose of study agent
* Donation or loss of ≥ 1 unit of whole blood or plasma within 2 months prior to dosing
* History of severe allergic reactions or hypersensitivity
* Current or former smoker with a smoking history of ≥10 pack-years
* Receipt of immunosuppressant therapies or biologic therapy for asthma within 6 months of screening
* Other investigational agent(s) within 30 days of dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence, nature, and severity of serious adverse events (SAEs) with a single dose of PRA-216 in healthy volunteers (SAD arm) | Up to 25 weeks
  Incidence, nature, and severity of serious adverse events (SAEs)
Phase 1: Incidence, nature, and severity of serious adverse events (SAEs) of multiple doses of PRA-216 in healthy volunteers (MAD arm) | up to 29 weeks
  Incidence, nature, and severity of and serious adverse events (SAEs)
Phase 2a: To evaluate the effect of multiple doses of PRA-216 compared to placebo on exhaled nitric oxide (FeNO) in asthma participants | Up to 29 weeks
  Fractional exhaled nitric oxide (FeNO) is a non-invasive biomarker of airway inflammation in asthma.

SECONDARY OUTCOMES:
Phase 1: Immunogenicity of PRA-216: ADA in healthy volunteers | Up to 29 weeks
  Incidence and magnitude of anti-drug antibody following single or multiple doses of PRA-216
Phase 1: Pharmacokinetics of PRA-216: Tmax in healthy volunteers | Up to 29 weeks
  Time to maximum concentration of drug in plasma following single or multiple doses of PRA-216
Phase 1: Pharmacokinetics of PRA-216: AUC in healthy volunteers | Up to 29 weeks
  Area under the curve following single or multiple doses of PRA-216
Phase 1: Pharmacokinetics of PRA-216: Cmax in healthy volunteers | Up to 29 weeks
  Maximum concentration of PRA-216 in plasma following single or multiple doses of PRA-216.
Phase 2a: Incidence, nature, and severity of serious adverse events (SAEs) of PRA-216 in patients with asthma | Up to 29 weeks
  Incidence, nature, and severity of serious adverse events (SAEs)
Phase 2a: Immunogenicity of PRA-216: ADA in patients with asthma | Up to 29 weeks
  Incidence and magnitude of anti-drug antibody following drug administration
Phase 2a: Pharmacokinetics of PRA-216: Tmax in patients with asthma | Up to 29 weeks
  Time to maximum concentration of drug in plasma following multiple doses of PRA-216
Phase 2a: Pharmacokinetics of PRA-216: AUC in patients with asthma | Up to 29 weeks
  Area under the curve of PRA-216 following multiple doses of PRA-216
Phase 2a: Pharmacokinetics of PRA-216: Cmax in patients with asthma | Up to 29 weeks
  Maximum concentration in plasma of PRA-216 following multiple doses

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Linear, Joondalup, Western Australia
  - Linear, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No